CLINICAL TRIAL: NCT05907928
Title: Radiographic Evaluation of Adaptation of New Radio-opaque Universal Adhesive Compared to Universal Adhesive in Proximal Restorations: Randomized Clinical Trial
Brief Title: Radiographic Evaluation of Adaptation of Universal Adhesives
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Associate Professor, Department of Conservative Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Universal adhesive plus
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Class II Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radio-opaque universal adhesive (Experimental): Radio-opaque universal adhesive
  Interventions: Other: Scotchbond universal adhesive plus
- Conventional universal adhesive (Active Comparator): Conventional universal adhesive
  Interventions: Other: Single bond Universal

INTERVENTIONS:
Other: Scotchbond universal adhesive plus — New generation BPA free universal adhesive
  Arms: Radio-opaque universal adhesive
Other: Single bond Universal — Radiolucent universal adhesive
  Other Names: Scotchbond universal adhesive
  Arms: Conventional universal adhesive

SUMMARY:
Class 2 restorations are analyzed to see whether or not the use of modified universal adhesive will result in similar adaptation to conventional universal adhesive.

DETAILED DESCRIPTION:
The newly modified adhesive with its careful formulation offers:

Radiopacity like dentin to reduce the risk of X-ray misdiagnosis and overtreatment. Ability to bond and seal caries-affected dentin to support minimally invasive preparation guidelines and maximize preservation of natural tooth structure. Adhesion to all dental substrates and all direct and indirect materials, including glass ceramics. Full dual- and self-cure compatibility without the need for an additional dual-cure activator bottle. A bisphenol A (BPA) derivative-free formulation to alleviate concerns about BPA in dental materials. A fully aligned system with RelyX™ Universal Resin Cement, offering excellent bond strength for virtually all dual-cure resin cement indications.

As with any new material or technique, clinical evaluations are needed to demonstrate the value of universal bonding agents adequately. Therefore, the aim of the current study was to evaluate adaptation of class 2 restorations either using radio-opaque universal adhesive or universal adhesive using digital radiography.

ELIGIBILITY:
Inclusion Criteria:

* Small to moderate carious proximal lesions. (International caries detection and assessment system (ICDAS) scores 3,4)
* Good oral hygiene (mild to moderate plaque accumulation)
* Vital teeth with no signs of irreversible pulpitis.
* Presence of favorable occlusion and normal contact with adjacent teeth.

Exclusion Criteria:

* Patients with systemic diseases, severe medical complications or allergic history concerning methacrylates.
* Lack of patient compliance, pregnancy, rampant caries, heavy smoking or xerostomia.
* Evidence of parafunctional habits and tempromandibular joint disorders.
* Deep carious defects (close to pulp, less than 1 mm distance).
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Endodontically treated teeth.
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism.
* Severe periodontal affection.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment of adaptation of restoration | 1week
  Modified USPHS criteria: Score A : harmonious transition between restoration and tooth; Score B: Presence of adhesive line (Radiolucent zone) below the restoration

CONTACTS AND LOCATIONS:
Overall Officials: Omar Shaalan, PhD, Principal Investigator — Lecturer, Department of Conservative Dentistry
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No